CLINICAL TRIAL: NCT03749174
Title: Radius Fracture Anesthesia and Rehabilitation (RADAR)
Acronym: RADAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgård, Associate professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RADAR
Record Dates: First submitted 2018-08-22; First posted 2018-11-21 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Radial Fracture
Keywords: Radial fracture; Anesthetic; Plaster; Cast; Orthosis; Brace; Postoperative pain; Quality of Recovery
MeSH Terms: conditions — Radius Fractures; Pain, Postoperative | interventions — Orthotic Devices; Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Patients are subdivided into 3 groups where one group is further subdivided into 2 groups
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Long acting anesthetic block/plaster (Active Comparator): Intervention 1: Blockade will be given supraclavicularly with Long acting local Anesthetic (n=30) combined with post operative plaster immobilization.
  Interventions: Procedure: Long acting Supraclivicular block vs Short acting Supraclavicular block
- Short acting anesthetic block/plaster (Active Comparator): Intervention 2: Blockade will be given supraclavicularly with Short acting local anesthetic (n=30) combined with plaster immobilisation postoperatively
  Interventions: Procedure: Long acting Supraclivicular block vs Short acting Supraclavicular block
- Short acting anesthetic block/orthotic (Active Comparator): Intervention 3: Blockade will be given supraclavicularly with Short acting local anesthetic (n=30) and combined with orthosis for postoperative immobilisation
  Interventions: Procedure: Long acting Supraclivicular block vs Short acting Supraclavicular block
- General Anesthesia and plaster (Active Comparator): Intervention 4: General anesthesia wil be administered for surgical procedure combined with postoperative plaster immobilisation (n=30),
  Interventions: Procedure: Long acting Supraclivicular block vs Short acting Supraclavicular block

INTERVENTIONS:
Procedure: Long acting Supraclivicular block vs Short acting Supraclavicular block — Patients are randomized to receive; long-acting Supraclavicular plexus block or short-acting Supraclavicular plexus block or general anesthesia
  Sub group randomized to plaster/cast or orthosis/brace, both having short-acting block
  Other Names: Long acting anesthetic block/plaster; Short acting anesthetic block/plaster; Short acting anesthetic block/orthosis; General Anesthesia and plaster

SUMMARY:
Distal fracture of the radial bone is the commonest fracture and is also connected to osteoporosis. Normally the operation is performed under neuroaxial blockade and sedation. When the blockade rapidly vanish many patients experience a rebound pain much severer that than the actual trauma pain. If long acting local anesthetics are used this will occur during night time and many patients will go to the emergency room for pain treatment. Short acting local anesthetics may make it possible to treat patients pain in-house prior to leaving the hospital. In this study

DETAILED DESCRIPTION:
This investigation is a joint study involving Occupational Therapist, Orthopedic surgeons and Anesthesiologist. Distal fracture of the radial bone is the commonest fracture, mainly in elder females with osteoporosis and also obesity. Normally 75% of patients are treated with plaster after fracture repositioning. The remaining 25% are operated upon. Routinely, the operation is performed under neuroaxial blockade and sedation. When the blockade rapidly vanish many patients experience a rebound pain much severer than the initial trauma pain. If long acting local anesthetics are used the blockade will be terminated during night and many patients will go to the Emergency room for pain treatment. Short acting local anesthetics may make it possible to treat patients pain in-house prior to hospital discharge and thus reduce severe rebound pain.

In this study patients with radial fractures are included and operated upon by a standard surgical operation with plate and screws. They will receive either 1) ultra sound guided supraclavicular block long-acting (n=30) local anesthetic , 2) ultra sound guided supraclavicular block short-acing (n=60) local anesthetics or 3) general anesthesia (n=30) to provide analgesia during the operational procedure. Patients given an ultra sound guided blockade with short-acting local anesthetic (n=60) are further sub-divided into receiving either postoperative plaster/cast (n=30) or an orthosis/brace (n=30).

Patients pain will be measured by Numeric Rating scale (0 = no pain and 10 worst possible pain) during the first 7 postoperative days. The opioid consumption will be noted by personal contact intermittently by telephone and by a pain diary until day 7. Both parametric and none-parametric analysis will be conducted.

Quality of recovery will be assessed by Quality of Recovery Scale 15 at 5 occasions. Adverse effects and unplanned health care contacts will also be gathered.

After 3 days the Occupational Therapist will control the patients followed by investigations at 2, 6 12 and 52 weeks. The patients will be graded the Patient rated Wrist Evaluation (PRWE) and Michigan Outcomes Questionnaire (MHQ) Edema will be measured and strength will be measured by Jamar dynamometer, Finally, Sense of coherence will be measured by KASAM-13

ELIGIBILITY:
Inclusion Criteria:

* Understands native language
* Cognitive intact
* Fracture types AO 23..A and AO 23.C.1
* Operated within 18 days from initial trauma

Exclusion Criteria:

* Not fulfilling inclusion criterias
* High energy trauma
* Ligament injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Rebound pain, difference in pain (NRS) at rest at 24-hours and further during the first three days after surgery between short acting block (mepivacaine) and long acting block (ropivacaine), with General Anesthesia being control group. | 72 hours
  Postoperative pain measured by numeric pain rating scale (NRS), where 0 = no pain and 10 = worst possible pain.
Quality of Recovery; difference in sum median and its five domains of QoR-15 score at baseline, 24 hours, 72 hours and 7 days after surgery between the two groups cast and orthosis/brace. - Anesthesiology part 2 | 1st three postoperative days
  Quality of Recovery scale 15 assessment
Post surgery arm function - Occupational therapist | 12 months
  Influence of immobilization by plaster or orthosis/brace

SECONDARY OUTCOMES:
Post surgery opioid requirement - Anesthesiology part | day 1 to 3 after surgery, including day 7 assessing immobilization (cast/brace)
  daily opioid requirement mg dose
Perioperative time events - Anesthesiology part | perioperatively
  Perioperative time events; e.g. duration of surgery, anesthesia, Theatre time and recovery room stay
Postoperative Nausea and Vomiting - Anesthesiology part | up to 72 hours post surgery
  Any experience of PONV
Unplanned health care contact - Anesthesiology part | 1st postoperative week
  any unplanned contact with health care, emergency department visit, phone calls, GP visits etc.
Post surgery arm status 1 - Occupational therapist | 12 months
  Clinical evaluation of post surgery arm status by a physiotherapist including: oedema,
Post surgery arm status 2 - Occupational therapist | 12 months
  Clinical evaluation of post surgery arm status by a physiotherapist including: grip strength
Post surgery arm status 3 - Occupational therapist | 12 months
  Clinical evaluation of post surgery arm status by a physiotherapist including sense of coherence.

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Nellgard, MD PhD, Principal Investigator — Göteborg University
Locations (1):
- SahlgrenskaUH, Mölndal, VGR, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galos DK, Taormina DP, Crespo A, Ding DY, Sapienza A, Jain S, Tejwani NC. Does Brachial Plexus Blockade Result in Improved Pain Scores After Distal Radius Fracture Fixation? A Randomized Trial. Clin Orthop Relat Res. 2016 May;474(5):1247-54. doi: 10.1007/s11999-016-4735-1. Epub 2016 Feb 11. PMID 26869374
- [Derived] Sellbrant I, Karlsson J, Jakobsson JG, Nellgard B. Supraclavicular block with Mepivacaine vs Ropivacaine, their impact on postoperative pain: a prospective randomised study. BMC Anesthesiol. 2021 Nov 9;21(1):273. doi: 10.1186/s12871-021-01499-z. PMID 34753423